CLINICAL TRIAL: NCT01850095
Title: The Influence of Peripheral Androgen Conversion at Toll-like Receptors-2 and CD1d Expressions in Human Keratinocytes as Well as Their Modulation After 6 Months Treatment With Oral Contraceptive.
Brief Title: The Influence of Peripheral Androgen Conversion at Women Adult Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marco Alexandre Dias da Rocha (Other)
Collaborators: Fleury (Unknown); Associacao Fundo de Incentivo a Psicofarmcologia (Other); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Marco Alexandre Dias da Rocha, MD, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1622/11
Record Dates: First submitted 2013-05-01; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Acne; Quality of Life
Keywords: acne; adult; women; TLR; CD1d; androgens
MeSH Terms: conditions — Acne Vulgaris | interventions — azelaic acid; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- treatment 1 (Active Comparator): topical acid azelaic, used 2 times a day for 6 months
  Interventions: Drug: treatment azelaic acid (azelan)
- treatment 2 (Active Comparator): contraceptive with drospirenone/ethinyl estradiol used for 6 months
  Interventions: Drug: dorspirenone/ethynil estradiol
- control (No Intervention): control group ( only take biopsies and blood samples )

INTERVENTIONS:
Drug: treatment azelaic acid (azelan) — treatment for 6 months
  Other Names: azelaic acid (azelan)
  Arms: treatment 1
Drug: dorspirenone/ethynil estradiol
  Other Names: (yaz)
  Arms: treatment 2

SUMMARY:
Acne vulgaris is a chronic inflammatory disease that affects the pilosebaceous unit. Recent studies have demonstrated an increase number of acne cases in adult women. These cases are predominantly normoandrogenic and have some clinical differences when compared with the most common group, the adolescent. The local glandular metabolism converts some hormonal precursors to more active substances that increase the sebum production, leaving these areas more prone to increase the colonization to Propionibacterium Acnes (P. Acnes). Toll-like receptor 2, expressed by inflammatory cells play a crucial role in the innate immune response to this bacterium. Previous studies confirm that exist a reduced expression of CD1d by keratinocytes in acne lesion, what can be interpreted as a low antigen-present function. The influence of hormonal alteration in the sebaceous glands could modulate the expressions of TLR-2 and CD1d explaining the persistence of lesions in adult women. The change to more estrogenic metabolism, with use of specific contraceptive pills could normalize this immune-mediated inflammatory process.

Objective

To analyze how the peripheral androgen conversion can influence the toll-like receptor 2 and CD1d expression in women with inflammatory acne before and after 6 months of oral contraceptives with anti-androgen activity.

ELIGIBILITY:
Inclusion Criteria:

To all:

1. Signing the consent form before any study procedures;
2. women aged 26 to 44 years, not pregnant and in good health;
3. no topical treatment for acne in the past three months,
4. absence of the use of oral antibiotics in the last 3 months;
5. absence of the use of isotretinoin in the last 2 years;
6. absence of oral contraceptive use in the last 3 months;
7. absence of clinical evidence of immunosuppression and
8. accordance with the conditions of study, ability to understand and strictly follow the instructions given.

For the oral contraceptives group:

1. No contraindications to the use hormonal contraceptives.

For the azelaic acid group:

1. Absence of hypersensitivity to azelaic acid.

Exclusion Criteria:

For all

1. Women who do not agree with the conditions of the study or without the ability to understand and closely follow the guidelines received without availability to attend the revaluations or who refuse to sign the Informed Consent Form;
2. pregnant or lactating women;
3. use of the following oral medications: cortisone derivatives, lithium, anticonvulsants, isoniazid, oral contraceptives, androgens, danazol, iodides, bromides, disulfiram, cyclosporine, azathioprine, thiuram, vitamins B2, B6 and B12;
4. treatment of facial skin with topical retinoids (tretinoin and adapalene), azelaic acid, benzoyl peroxide, clindamycin, erythromycin, nicotinamina, alone or in combination, in the past 3 months;
5. treatment with oral antibiotics in the past 3 months;
6. acnogenics cosmetics.

For the group treated with oral contraceptives:

1. Presence of contraindications to oral contraceptive use:

1. Smokers over 35 years;
2. history of deep venous thrombosis;
3. history of stroke;
4. history of breast cancer;
5. presence of jaundice, and severe active liver disease or biliary disease;
6. diabetes mellitus for more than 20 years or eye injury, or neurological impairment;
7. blood pressure greater than or equal to 160 to 100 for systolic and diastolic;
8. cardiovascular disease and
9. presence of severe headache associated with blurred vision frequently.

For the group treated with azelaic acid:

1.Presense of allergic and / or irritating symptoms to the use of azelaic acid.

For the control group 1:

1. History, clinical signs and / or laboratory evidence of hyperandrogenism. 2 .Presence of inflammatory acne.

-

Ages: 26 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of the treatment group | 6 months
  by the researcher: by counting the inflammatory lesions. by the research subjects: the general appearance of skin at the time of study entry and after the treatment. Will be used a 4-point scale: 0 = no acne, 1 = mild acne, moderate acne, and 2 = 4 = severe acne.

SECONDARY OUTCOMES:
Photographic study of the treatment group | 6 months
  This evaluation will be performed by two independent dermatologists, the degree of change in the intensity of acne, comparing the pre and post treatment photos through a 5-point scale: -2 = much worse, -1 = worse, 0 = unchanged; +1 = better, +2 = much better.

OTHER OUTCOMES:
Application of the questionnaire index of quality of life in Acne | 6 months
  AcneQol (Girman et al, 1996, Martin et al, 2001, Fehnel et al, 2003),
Immunohistochemical analysis with quantitative digital blind: | 6 months
  For immunohistochemistry will be used the following markers:
  * a polyclonal rabbit anti-TLR2 (ABBIOTEC 251,110) Biogen, Brazil.
  * mouse monoclonal anti-CD1d, clone NOR3.2 (Genway 20-272-1903). Biogen, Brazil.
  Statistical comparisons are made between the following groups: control group 2 and the region with inflammatory lesions in the treatment group, region and region inflammatory non-inflammatory group of medications and treatment before inflammatory region before and after treatment.
Serological blood measurements | 6 months
  Comparison of serological blood measurements of free and total testosterone, dihydroepiandrosterone sulfate (DHEAS), luteinizing hormone (LH), follicle-stimulating hormone (FSH), and androsterone glucuronide, before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: marco rocha, md, Principal Investigator — UNIFESP-EPM
Locations (1):
- Federal University of São Paulo-Dermatology, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Bhambri S, Del Rosso JQ, Bhambri A. Pathogenesis of acne vulgaris: recent advances. J Drugs Dermatol. 2009 Jul;8(7):615-8. PMID 19588637
- [Background] Shen Y, Wang T, Zhou C, Wang X, Ding X, Tian S, Liu Y, Peng G, Xue S, Zhou J, Wang R, Meng X, Pei G, Bai Y, Liu Q, Li H, Zhang J. Prevalence of acne vulgaris in Chinese adolescents and adults: a community-based study of 17,345 subjects in six cities. Acta Derm Venereol. 2012 Jan;92(1):40-4. doi: 10.2340/00015555-1164. PMID 21710106
- [Background] Gollnick H, Cunliffe W, Berson D, Dreno B, Finlay A, Leyden JJ, Shalita AR, Thiboutot D; Global Alliance to Improve Outcomes in Acne. Management of acne: a report from a Global Alliance to Improve Outcomes in Acne. J Am Acad Dermatol. 2003 Jul;49(1 Suppl):S1-37. doi: 10.1067/mjd.2003.618. No abstract available. PMID 12833004
- [Background] Thiboutot D. Acne: hormonal concepts and therapy. Clin Dermatol. 2004 Sep-Oct;22(5):419-28. doi: 10.1016/j.clindermatol.2004.03.010. PMID 15556729
- [Background] Kurokawa I, Danby FW, Ju Q, Wang X, Xiang LF, Xia L, Chen W, Nagy I, Picardo M, Suh DH, Ganceviciene R, Schagen S, Tsatsou F, Zouboulis CC. New developments in our understanding of acne pathogenesis and treatment. Exp Dermatol. 2009 Oct;18(10):821-32. doi: 10.1111/j.1600-0625.2009.00890.x. Epub 2009 Jun 23. PMID 19555434
- [Background] White GM. Recent findings in the epidemiologic evidence, classification, and subtypes of acne vulgaris. J Am Acad Dermatol. 1998 Aug;39(2 Pt 3):S34-7. doi: 10.1016/s0190-9622(98)70442-6. PMID 9703121
- [Background] Goulden V, Stables GI, Cunliffe WJ. Prevalence of facial acne in adults. J Am Acad Dermatol. 1999 Oct;41(4):577-80. PMID 10495379
- [Background] Goulden V, Clark SM, Cunliffe WJ. Post-adolescent acne: a review of clinical features. Br J Dermatol. 1997 Jan;136(1):66-70. PMID 9039297
- [Background] Poli F, Dreno B, Verschoore M. An epidemiological study of acne in female adults: results of a survey conducted in France. J Eur Acad Dermatol Venereol. 2001 Nov;15(6):541-5. doi: 10.1046/j.1468-3083.2001.00357.x. PMID 11843213